CLINICAL TRIAL: NCT06582173
Title: Mapping the Healthcare Pathway to Specialised Multidisciplinary Assessment of 12-25 Year Olds With Somatic Symptom Disorder: a Monocentric Descriptive Study Based on Interviews Assisted by a Biographical Grid
Brief Title: Mapping the Healthcare Pathway to Multidisciplinary Assessment of 12-25 Year Olds With Somatic Symptom Disorder
Acronym: PSOMA
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240890; 2024-A01371-46 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Somatic Symptoms; Medically Unexplained Symptoms; Somatoform Disorders
Keywords: Somatic symptoms; Somatoform disorder; Medically unexplained symptoms; Healthcare pathway; Healthcare trajectory; Care episodes; Health Care Utilization; Adolescent; Young Adult
MeSH Terms: conditions — Medically Unexplained Symptoms; Somatoform Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adolescents: Patients aged 12 to 25 years old and diagnosed with SSD by a specialised multidisciplinary team
  Interventions: Other: Face-to-face interviews assisted by a biographical grid
- Parents: Parents of an adolescent included
  Interventions: Other: Face-to-face interviews assisted by a biographical grid

INTERVENTIONS:
Other: Face-to-face interviews assisted by a biographical grid — Face-to-face interviews assisted by a biographical grid.
  Healthcare event of the adolescent :
  * medical specialist appointment
  * general practitioner appointment
  * emergency services use
  * hospital admission
  * diagnostic test
  * medication use
  * non-pharmacological treatment
  * nursing or physical therapy
  * alternative care
  Biographical of the adolescent :
  * Education event
    * Class/level
    * School
    * Attendance
    * Special arrangements
    * Grades
    * Off school education
  * Family event
    * Separation/union
    * Birth/death
    * Leave/Arrival
    * Location/Moving
    * Disease/accident
  * Peer events
    * Friendships
    * Love interests
    * Bullying
  * Leisure & interests events
    * Activity
    * Frequency

SUMMARY:
This study aims to describe the course of successive care events that follow individuals with somatic symptom disorder until they are assessed by a specialized multidisciplinary team. Data is collected during interviews with subjects aged 12 to 25 years old accompanied by their parents. A biographical grid is used to retrospectively identify all care events that occurred from first symptoms until multidisciplinary assessment. Life events and symptoms are collected as well to explore how history of healthcare consumption is linked to other trajectories. A qualitative analysis of the recorded interviews aims to describe the subjective experience of this healthcare pathway.

DETAILED DESCRIPTION:
Somatic symptom disorders (SSD), previously labelled Somatoform disorders, are known to challenge healthcare professionals and systems, as those common conditions reducing quality of life often lead to excessive referrals and investigations before adequate diagnosis and management. Although studies have proved multiple interventions to be effective and cost-effective in various clinical settings, little is known about the accurate healthcare utilization associated with SSD. Such analysis faces the complexity of SSD detection and labelling due to heterogeneous clinical presentations and disputed cross-disciplinary classifications. Even though healthcare is known to be a core theme of patient experience of SSD, the investigators lack data describing the trajectory of care and the expectations, perceived help and triggering events associated with healthcare services use. A better understanding of the healthcare pathway those patients follow will help implement evidence-based treatment effectively.

The aim of this study is to trace back the pathway of care that individuals follow before they eventually undergo a specialised multidisciplinary assessment.

This descriptive study relies on data retrospectively collected from patients and their parents during face-to-face interviews assisted by a biographical grid. Inclusion criteria for patients are to be aged 12 to 25 years old and to be diagnosed with SSD by a specialised multidisciplinary team. Variables measured to describe the healthcare pathway are chosen according to professional experience and literature review. They are collected alongside concomitant life events both to reduce memory bias and to explore determinants and effects of healthcare consumption as a secondary outcome. The subjective experience of this healthcare pathway described by patients and their parents is analysed qualitatively in the verbatim of the audio recorded interview.

ELIGIBILITY:
Inclusion Criteria:

Criteria relating to the population studied:

* Age between 12 and 25 years old
* Diagnosis of somatic symptom disorder and derivatives (DSM 5) after specialized multidisciplinary evaluation by the team of the Maison des Adolescents of Cochin hospital (Maison de Solenn).

Criteria relating to the additional population participating in the research:

- Being a parent of a subject who has received the diagnosis of somatic symptom disorder and derivatives (DSM 5) after specialized multidisciplinary evaluation at the Maison des Adolescents of Cochin Hospital (Maison de Solenn).

Exclusion Criteria:

Criteria relating to the population studied:

* Age less than 12 years or greater than 25 years at the time of assessment,
* Subject presenting ongoing psychiatric decompensation, that is to say a state of mental health breaking with their baseline state and requiring rapid care which does not allow a research interview to be carried out.

Criteria relating to the additional population participating in the research:

None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are selected among patients assessed in the recruiting centre, whatever their course after assessment.
  The recruiting centre is an adolescent clinic which is part of a public teaching hospital in Paris, France. The centre provides inpatient and outpatient care delivered by a multidisciplinary team. Patients aged 11 to 18 can be referred to this centre by a healthcare professional or can directly access to care, regardless of their living area.
  For each patient included, parents are asked to participate to research interviews to help map the healthcare pathway their child followed.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of healthcare events | Day of inclusion
  Successive healthcare events of individuals with somatic symptom disorder, from first symptoms to specialised multidisciplinary assessment

SECONDARY OUTCOMES:
Raise of healthcare events occurrence | Day of inclusion
  Raise of healthcare events occurrence following the occurrence of somatic symptoms.
  From first symptoms to specialised multidisciplinary assessment
Raise of life events occurrence | Day of inclusion
  From first symptoms to specialised multidisciplinary assessment
Decrease of healthcare events occurrence | Day of inclusion
  Decrease of healthcare events occurrence following the occurrence of somatic symptoms.
  From first symptoms to specialised multidisciplinary assessment
Decrease of life events occurrence | Day of inclusion
  From first symptoms to specialised multidisciplinary assessment
Modification of somatic symptoms occurrence | Day of inclusion
  From first symptoms to specialised multidisciplinary assessment
Modification of life events occurrence | Day of inclusion
  Modification of life events occurrence following healthcare. From first symptoms to specialised multidisciplinary assessment
Qualitative analysis of the transcribed interviews | Up to 24 months
  Identification of themes emerging from the qualitative analysis of the transcribed interviews

CONTACTS AND LOCATIONS:
Overall Officials: Maude LUDOT-GREGOIRE, MD, PhD, Principal Investigator — Maison des Adolescents - Cochin Hospital - AP-HP
Locations (1):
- Maison de Solenn Maison des Adolescents, Cochin Hospital, Paris, IDF, France

REFERENCES:
- [Background] Joustra ML, Janssens KA, Bultmann U, Rosmalen JG. Functional limitations in functional somatic syndromes and well-defined medical diseases. Results from the general population cohort LifeLines. J Psychosom Res. 2015 Aug;79(2):94-9. doi: 10.1016/j.jpsychores.2015.05.004. Epub 2015 May 16. PMID 26026696
- [Background] van Dessel N, den Boeft M, van der Wouden JC, Kleinstauber M, Leone SS, Terluin B, Numans ME, van der Horst HE, van Marwijk H. Non-pharmacological interventions for somatoform disorders and medically unexplained physical symptoms (MUPS) in adults. Cochrane Database Syst Rev. 2014 Nov 1;2014(11):CD011142. doi: 10.1002/14651858.CD011142.pub2. PMID 25362239
- [Background] Wortman MSH, Lokkerbol J, van der Wouden JC, Visser B, van der Horst HE, Olde Hartman TC. Cost-effectiveness of interventions for medically unexplained symptoms: A systematic review. PLoS One. 2018 Oct 15;13(10):e0205278. doi: 10.1371/journal.pone.0205278. eCollection 2018. PMID 30321193
- [Background] Gosselin A, Desgrees du Lou A, Lelievre E; PARCOURS Study Group. How to use sequence analysis for life course epidemiology? An example on HIV-positive Sub-Saharan migrants in France. J Epidemiol Community Health. 2018 Jun;72(6):507-512. doi: 10.1136/jech-2017-209739. Epub 2018 Feb 2. PMID 29437866
- [Background] Sawyer SM, Azzopardi PS, Wickremarathne D, Patton GC. The age of adolescence. Lancet Child Adolesc Health. 2018 Mar;2(3):223-228. doi: 10.1016/S2352-4642(18)30022-1. Epub 2018 Jan 30. PMID 30169257
- [Background] Kachaner A, Harim M, Combier A, Trouvin AP, Avouac J, Ranque B, Piot MA. Management perspectives from patients with fibromyalgia experiences with the healthcare pathway: a qualitative study. Front Med (Lausanne). 2023 Dec 1;10:1231951. doi: 10.3389/fmed.2023.1231951. eCollection 2023. PMID 38105901
- [Background] Hinton D, Kirk S. Families' and healthcare professionals' perceptions of healthcare services for children and young people with medically unexplained symptoms: a narrative review of the literature. Health Soc Care Community. 2016 Jan;24(1):12-26. doi: 10.1111/hsc.12184. Epub 2015 Feb 16. PMID 25684117
- [Background] Ludot M, Merlo M, Ibrahim N, Piot MA, Lefevre H, Carles ME, Harf A, Moro MR. ["Somatic symptom disorders" in adolescence. A systematic review of the recent literature]. Encephale. 2021 Dec;47(6):596-604. doi: 10.1016/j.encep.2021.04.007. Epub 2021 Sep 16. French. PMID 34538623